CLINICAL TRIAL: NCT00541853
Title: Comparison Between ARB and ARB Plus CCB on Incidence of Renal and Cardiovascular Events in Hypertensive ADPKD Patients
Brief Title: CCB Safety Study in Treatment of Hypertension of ADPKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyorin University (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADPKDCCB
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Kidney, Polycystic, Autosomal Dominant
Keywords: Autosomal Dominant Polycystic Kidney Disease; Hypertension; Angiotensin-2 Receptor Blocker; Calcium Channel Blocker; Kidney Volume
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Hypertension | interventions — candesartan; cilnidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): ADPKD patients with blood pressure above 130/85 are enrolled. The patients whose blood pressure is controlled under 130/85 by Candesartan alone are classified into group A.
  Interventions: Drug: Candesartan
- B (Experimental): The patients whose blood pressure is not controlled under 130/85 with ARB alone are randomized into group B or C. In group B, blood pressure is controlled by Candesartan plus Cilnidipine. If blood pressure is not lowered by Candesartan plus Cilnidipine alone, another antihypertensive agents except CCB and ACEI are allowable.
  Interventions: Drug: Candesartan and Cilnidipine
- C (Active Comparator): The patients whose blood pressure is not controlled under 130/85 with ARB alone are randomized into group B or C. In group C, blood pressure is controlled by Candesartan plus non-CCB agents such as beta- or alpha- adrenergic blockers or another ARB. Any CCB and ACEI are not allowable.
  Interventions: Drug: Candesartan plus non-CCB agents

INTERVENTIONS:
Drug: Candesartan — Candesartan upto 8mg
  Arms: A
Drug: Candesartan and Cilnidipine — Candesartan upto 8mg per day and Cilnidipine upto 20mg per day
  Arms: B
Drug: Candesartan plus non-CCB agents — Candesartan upto 8mg per day and other antihypertensive drugs except CCB and ACEI
  Arms: C

SUMMARY:
This study examines the safety and efficacy of calcium channel blocker (CCB) in the treatment of hypertension of Autosomal Dominant Polycystic Kidney Disease (ADPKD) patients. Angiotensin receptor blocker (ARB) was shown to have kidney protecting effects in patients with renal diseases including ADPKD, glomerulonephritis and diabetic nephropathy. In case whose blood pressure is not normalized by ARB alone, CCB is selected additionally. Recent research suggests genetic calcium channel disorder is responsible for the progression of ADPKD. It is not examined clinically if CCB treatment has any harmful effect to patients with ADPKD. This study examines the safety of Cilnidipine (CCB) in the ADPKD patients whose blood pressure is not controlled under 130/85 mmHg by Candesartan (ARB) alone.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients.
* Blood pressure measured at out-patient setting is above 130/85 mmHg.
* Age between 20 and 60 years old.
* Plasma creatinine less than 2.0mg in man and 1.5mg in woman.
* Patients give informed consent.

Exclusion Criteria:

* Patients with severe cardiovascular and hepatic disorders.
* Patients with complications of central nervous vascular disorders.
* Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods.
* Patients currently engaging in other experimental protocol.
* Patients with intracranial aneurysma.
* Patients who must use diuretics.
* Allergic patients to Candesartan or Cilnidipine.
* Patients whose hypertension is not controlled by medication of this protocol.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-12; Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Kidney Volume measured by MRI. | Every year

SECONDARY OUTCOMES:
Serum creatinine, hemodialysis, cardiovascular events and central nervous vascular events | any time during study period

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Higashihara, M.D., Study Chair — Kyorin University, School of Medicine
Locations (6):
- Japan (6):
  - Kyorin University School of Medicine, Mitaka, Tokyo
  - Department of Urology, National Hospital Organaization Chiba-East Hospital, Chiba, Chiba
  - Toranomon Hospital Kajigaya, Kidney center, Kanagawa
  - Toranomon Hospital, Kidney center, Tokyo
  - Division of Kidney and Hypertension, Department of Internal Medicine, Jikei University School of Medicine, Tokyo
  - Department of Urology, Teikyo University, School of Medicine, Tokyo

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Higashihara E, Nutahara K, Horie S, Muto S, Hosoya T, Hanaoka K, Tuchiya K, Kamura K, Takaichi K, Ubara Y, Itomura M, Hamazaki T. The effect of eicosapentaenoic acid on renal function and volume in patients with ADPKD. Nephrol Dial Transplant. 2008 Sep;23(9):2847-52. doi: 10.1093/ndt/gfn144. Epub 2008 Mar 27. PMID 18372389